CLINICAL TRIAL: NCT05661604
Title: Prospective Study to Investigate Acute Respiratory Virus Infections in Patients at High Risk for Severe Illness
Brief Title: A Study to Investigate Acute Respiratory Virus Infections in Participants at High Risk for Severe Illness
Acronym: BREEZE
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109291; NOPRODVIR0001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Viral Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, whole blood and nasosorption samples will be collected to retain DNA if required.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants at High Risk for Poor Outcomes From a Respiratory Infection: Data will be collected for participants at high risk for poor outcomes from a respiratory infection. The duration of participation per participant will be up to 12 months.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study to assess the incidence and key disease characteristics of symptomatic acute respiratory viral infections in a high-risk population at risk for poor outcomes. Duration of each participant will be up to 12 months.

SUMMARY:
The purpose of the study is to describe the rate of occurrence of clinical diagnosis of acute respiratory infection (an infection that affects normal breathing) and different types of respiratory pathogens (harmful organisms) of new respiratory infections in a population at high risk for severe illness.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent form (ICF) indicating understanding the purpose, procedures, and potential risks and benefits of the study, and is willing to participate in the study
* Participants at high risk for severe respiratory infections due to their immune-suppressive status and who fit in one or more of the following categories: a) Participants with hematologic malignancy (HM) including, but not limited to, acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), acute lymphoblastic leukemia (ALL), multiple myeloma (MM): i) Newly diagnosed, within 6 months of treatment initiation; including anticipation of cytotoxic and immunomodulatory therapy such as chimeric antigen receptor T (CAR-T) ii) Hematologic relapse within 6 months from anticipating treatment initiation for relapse iii) Participants with a history of HM who have maintained the immunosuppressive status in the opinion of the investigator and after consultation with the sponsor (that is, study responsible physician or scientists) b) Participants with a history of HM who have received hematopoietic cell transplant (HCT) within 1 year for autologous recipients or within 3 years for allogeneic recipients. c) Participants with a non-HM who have received HCT within 1 year for autologous recipients or within 3 years for allogeneic recipients. This can include, but is not limited to, participants who have received HCT due to lymphoproliferative disorders, solid tumors, primary immunodeficiency, bone marrow failure syndromes, hemoglobinopathies, sickle cell disease, or autoimmune disorders. d) Participants who have developed chronic graft vs host disease (GVHD) after HCT and are currently on immunosuppressive therapy
* Must be able to read, understand, and complete questionnaires
* Must be willing and able to connect current electronic health records from one or more providers

Exclusion Criteria:

* Has a clinical condition other than those specified in inclusion criterion 3 which, in the opinion of the investigator, could prevent, confound, or limit the protocol-specified assessments (for example, asthma and allergies)
* Is, in the opinion of the investigator, unlikely to adhere to the requirements of the study or is unlikely to complete the full course of observation
* Cannot communicate reliably with the investigator
* Has moderate-severe allergies that add complexity to the assessment of acute respiratory infection (ARI) episode
* Is currently enrolled in an interventional study that could interfere with the assessment of respiratory viral dynamics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at high risk for severe respiratory infections due to their immune-suppressive status.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Clinically Confirmed Acute Respiratory Infection (ARI) | Up to 1 year 3 months
  Number of participants with clinically confirmed ARI will be reported.
Number of Clinically Confirmed ARI Participants With Positive or Negative Infection Status for Each Respiratory Virus Tested | Up to 1 year 3 months
  Number of clinically confirmed ARI participants with positive or negative infection status for each respiratory virus tested will be reported.

SECONDARY OUTCOMES:
Number of Clinically Confirmed ARI Participants who Were Hospitalized | Up to 1 year 3 months
  Number of clinically confirmed ARI participants who were hospitalized will be reported.
Number of Clinically Confirmed ARI Participants who Experienced Complications | Up to 1 year 3 months
  Number of clinically confirmed ARI participants who experienced complications will be reported.
Number of Deaths in Clinically Confirmed ARI Participants | Up to 1 year 3 months
  Number of deaths in clinically confirmed ARI participants will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (3):
  - Stanford Hospital and Clinics, Palo Alto, California
  - Henry Ford Hospital, Detroit, Michigan
  - Fred Hutchinson Research Center, Seattle, Washington
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No